CLINICAL TRIAL: NCT07282275
Title: How Does Continued Use of Green Light Therapy Impact Outcomes?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Efforia, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 47409
Record Dates: First submitted 2025-12-05; First posted 2025-12-15 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Body Composition

STUDY DESIGN:
Intervention Model Description: Single Arm observational where participants act as their own control
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single arm where participants act as their own control (Experimental): Single Arm observational where participants act as their own control
  Interventions: Device: EmeraldLED

INTERVENTIONS:
Device: EmeraldLED — This device is a customizable, multi-wavelength therapeutic system designed for individualized cosmetic treatments. It features an easy-to-use interface with preprogrammed treatment categories, a wide pulsing frequency range from 1 to 15,000 Hz, and independent wavelength control for precise protocol tailoring. The system delivers five wavelengths-450 nm, 525 nm, 650 nm, 810 nm, and 980 nm-with an output power of 3,325 W and irradiance up to 119 mW/cm².
  The green light therapy provided in this study is set at 525 nm.

SUMMARY:
Already using Green Light Therapy? Explore how continued use with twice-weekly 20-minute sessions may continue to support positive changes in body composition. Discover whether this non-invasive wellness approach gets better over time to help support energy, balance, and renewal.

DETAILED DESCRIPTION:
This remotely administered decentralized trial is designed to meticulously investigate the effectiveness and potential benefits of green light therapy on body composition and overall well-being. As the wellness industry burgeons with claims of revolutionary treatments, the need for evidence-based research has never been more critical. Under the guidance of Ryan, the CEO of beem® Light Sauna, with an extensive background in the fitness and wellness industry, this study seeks to cut through the noise surrounding green light therapy. By leveraging the expansive network of beem®'s locations and their commitment to science-backed recovery modalities, this study aims to provide a robust evaluation of green light therapy's claims, focusing specifically on its impact on weight management and mood enhancement.

Participants in this study will engage in a series of green light therapy sessions, conducted entirely online to ensure convenience and broad accessibility. This innovative approach allows individuals from diverse geographical locations to partake in the study, enhancing the diversity of our participant pool and the generalizability of our findings. Throughout the study, participants will have their body composition meticulously analyzed, and their overall well-being assessed through scientifically validated measures, all from the comfort of their homes.

The primary objective of this investigation is to empower participants with tangible, personalized data concerning the effects of green light therapy on their health and wellness journey. By providing individualized feedback on changes in body composition and well-being, this study aims to illuminate the true efficacy of green light therapy. This endeavor not only seeks to validate or debunk existing claims but also to enrich the participant's understanding of their health, thereby enabling informed decisions regarding their wellness routines.

The significance of this study extends beyond the immediate benefits to the participants. By contributing to a pioneering exploration of green light therapy's potential in weight management and mood improvement, participants are at the forefront of a potentially transformative shift in health and wellness strategies. Although the study acknowledges limitations, including the necessity for subsequent comprehensive trials, the insights garnered here will pave the way for future health innovations. This trial stands as a beacon in the quest for truth, aiming to redefine approaches to weight management and wellness in an era increasingly focused on health consciousness.

ELIGIBILITY:
Inclusion Criteria:

* Can read and understand English.
* US resident.
* Willing and able to follow the requirements of the protocol.

Exclusion Criteria:

* Individuals with eye conditions
* Individuals not active with Green Light Therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2026-10-21 (Estimated); Study Completion 2026-10-21 (Estimated)

PRIMARY OUTCOMES:
Body Composition Measurement Form | Change from baseline (Day 1-3) in body composition at 4 weeks after the start of the intervention (Day 27-33).
  The Body Composition Measurement Form is specifically crafted to accurately track changes in body measurements relevant to individuals engaged in weight loss or bodybuilding. This form allows for the consistent recording of key physical metrics across various body parts, facilitating the evaluation of fitness progress. By using this form, individuals can obtain a clear picture of the physical changes resulting from their exercise routines and nutritional choices. Each measurement is to be recorded in centimeters to maintain uniformity and precision.
Quality of Life and Health Survey | Change from baseline (Day 1-3) in quality of life and health at 4 weeks after the start of the intervention (Day 27-33).
  This survey asks about your feelings towards your quality of life, health, and various areas of your life. It covers your experiences and feelings in the past four weeks. Please choose the answer that appears most appropriate.
Body Image and Self-Perception Survey | Change from baseline (Day 1-3) in body image and self-perception at 4 weeks after the start of the intervention (Day 27-33).
  This survey aims to understand an individual's perception of their body, attractiveness, and physical functionality. It contains multiple-choice questions with five options ranging from 'Strongly Disagree' to 'Strongly Agree'. The questions are divided into three categories: Body Satisfaction, Attractiveness Evaluation, and Physical Functionality Awareness.

CONTACTS AND LOCATIONS:
Locations (1):
- Efforia, New York, New York, United States

REFERENCES:
- See also: Additional information and join instructions on Efforia — https://app.efforia.com/wp-admin/admin.php?page=llms-course-builder&course_id=47374